CLINICAL TRIAL: NCT03568240
Title: Voice Acoustic Properties in People With OSAS (Obstructive Sleep Apnea Syndrome)
Brief Title: Voice Acoustic Properties in People With Obstructive Sleep Apnea Syndrome (OSAS)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0019-18-HYMC
Record Dates: First submitted 2018-05-30; First posted 2018-06-26 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 30 men suffering from apnea
  Interventions: Diagnostic Test: Patients suffering from Sleep apnea
- 15 men defined as snorers
  Interventions: Diagnostic Test: Patients suffering from Sleep apnea
- 15 men without complaints
  Interventions: Diagnostic Test: Patients suffering from Sleep apnea

INTERVENTIONS:
Diagnostic Test: Patients suffering from Sleep apnea — PSG test

SUMMARY:
The aim of this study is to examine whether voice acoustic properties has an influence on sleep apnea. Sleep apnea syndrome is defined as a sudden stop of more than ten seconds multiple times during sleep. The syndrome is common especially among men and occurs in 2%-4% of the population aged 30-60. The syndrome diagnosis is performed by an ENT (Ear, Nose and Throat) physician. The diagnosis is based on evaluation of anatomical structures in the sound path (nose and throat, jaw, pharynx and oral cavity) and a Polysomnography (PSG) test which quantifies the number and duration of breathing pauses during night sleep and additional parameters that monitor sleep. The syndrome has many negative consequences for those who suffer from it, including fatigue , lack of concentration, hypertension, diabetes ,heart disease, stroke and even death. Therefore, early diagnosis is important.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older men who meet the criteria for disorders such as apnea.
* 18 years old men and older who meet the criteria of snores based on screening questionnaires.
* 18 years old men and older who don't suffer from disorders such as apnea and do not suffer from snoring.

Exclusion Criteria:

* Smoking Patients or smoked in the past.
* Having neurological disorders.
* Having swallowing trouble.
* Having Respiratory problems.
* Having Neuroendocrine problems.
* Having Voice disorders.
* Patients who were previously head or/and neck operated

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 men patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Compare differences in acoustic properties of phonetics i,a,u, n,m | half hour
  Subjects will be recorded in a variety of positions expressing the phonetics i,a,u, n,m. and the results will be documented and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Itzhak Braverman, MD, Principal Investigator — Hillel Yaffe Medical Center

IPD SHARING:
Plan to Share IPD: No